CLINICAL TRIAL: NCT01209962
Title: A Pilot Study of Diffusion MRI in the Assessment of Pancreatic Tumor Response
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2008.034; HUM 20979 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2010-04-02; First posted 2010-09-27 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort: The majority of recruited patients will be treated on protocol HUM00004531 "A Multi-Institutional Phase II Study of Neoadjuvant Gemcitabine and Oxaliplatin with Radiation Therapy in Patients with Pancreatic Cancer".

SUMMARY:
Patients with pancreatic cancer are treated with combinations of surgery, radiation therapy and chemotherapy, depending on the location of the cancer and other individual patient health factors. The goals of therapy are to reduce or eliminate the cancer cells, but without serious damage to normal cells. Investigators at The University of Michigan are conducting a research project, to see if treatment effects on an individual patient's cancer cells can be detected early by new imaging tests in patients with resectable pancreatic cancer undergoing neoadjuvant chemoradiotherapy.

DETAILED DESCRIPTION:
Patients with pancreatic cancer are treated with combinations of surgery, radiation therapy and chemotherapy, depending on the location of the cancer and other individual patient health factors. The goals of therapy are to reduce or eliminate the cancer cells, but without serious damage to normal cells.Each patient is unique in terms of the cancer type and location and its sensitivity to treatments. Investigators at The University of Michigan are conducting a research project to see if treatment effects on an individual patient's cancer cells can be detected early by new imaging tests in patients with resectable pancreatic cancer undergoing neoadjuvant chemoradiotherapy. Each patient is unique in terms of the cancer type and location and its sensitivity to treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic or cytologic proof of pancreatic cancer, for whom the treatment plan, at the time of enrollment, is neoadjuvant chemoradiotherapy followed by surgical resection.
* Patients must be >18 years old.
* Patients cannot weight over 300 pounds, the weight limit of the MRI table.
* Patients must have adequate renal function (estimated glomerular filtration rate > 60 mL/min/m2), to minimize the small risk of nephrogenic systemic sclerosis associated with gadolinium injection.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of UM hospital.

Exclusion Criteria:

* Patients must have no previous radiation to the abdomen.
* Patients who are pregnant or lactating are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologic or cytologic proof of pancreatic cancer, for whom the treatment plan, at the time of enrollment, is neoadjuvant chemoradiotherapy followed by surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2015-05-26 (Actual); Study Completion 2015-05-26 (Actual)

PRIMARY OUTCOMES:
Diffusion MRI | 5 years
  The goal is to develop a functional imaging method that would be a better predictor of pathological response than the current CT standard. Diffusion MRI has the potential to measure early cellular changes that occur in response to successful therapies, such as chemoradiation, and has been demonstrated to be an early predictor not only of therapeutic response, but also of overall survival for other malignancies.

SECONDARY OUTCOMES:
Apparent Diffusion Coefficient (ADC) | 5 years
  Demonstrate that the distribution of Apparent Diffusion Coefficient in pancreatic tumors, as measured by diffusion MRI, changes in response to neoadjuvant chemoradiotherapy, and characterize the differences in the distributions between histopathologic responders and non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Cuneo, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States